CLINICAL TRIAL: NCT02015260
Title: A Randomised, Multicentre, Double-blind, Placebo-controlled, Dose-ranging Trial to Evaluate the Efficacy, Safety and Tolerability of Three Dose Regimens of Topical Nitric Oxide in Patients With Anogenital Warts
Brief Title: A Trial of the Efficacy and Safety of Topical Nitric Oxide in Patients With Anogenital Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANA/2/C
Record Dates: First submitted 2013-08-06; First posted 2013-12-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2013-12

CONDITIONS: Anogenital Warts; Condylomata Acuminata
Keywords: human papilloma virus infection; Anogenital warts; condylomata acuminata
MeSH Terms: conditions — Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): placebo 0% nitrite cream and placebo 0% citric acid cream
  Interventions: Drug: Placebo
- Topical NO Dose A (Active Comparator): 3% sodium nitrite + 4.5% citric acid twice daily
  Interventions: Drug: Topical NO
- Topical NO Dose B (Active Comparator): 6% sodium nitrite + 9% citric acid once daily
  Interventions: Drug: Topical NO
- Topical NO Dose C (Active Comparator): 6% sodium nitrite + 9% citric acid twice daily
  Interventions: Drug: Topical NO

INTERVENTIONS:
Drug: Topical NO — Varying doses of sodium nitrite and citric acid co-applied to warts
  Other Names: Acidified Nitrite vs Placebo
  Arms: Topical NO Dose A; Topical NO Dose B; Topical NO Dose C
Drug: Placebo — Placebo
  Other Names: Placebo nitrite cream and placebo citric acid cream
  Arms: placebo

SUMMARY:
Objective To assess the efficacy of the topical application of Nitric Oxide, delivered using acidified nitrite.

Design Multicentre, randomized, controlled, dose ranging trial. A control arm and three doses of acidified nitrite applied topically for 12 weeks with a further 12 weeks of follow up.

Setting The trial setting was in European genitourinary medicine clinics

Participants Male and female volunteers over 18 years of age with between 2 and 50 ano-genital warts, 328 were screened for eligibility and 299 subjects from 40 centres were randomised.

Exclusions Pregnancy; concomitant Sexually Transmitted Disease; internal warts requiring treatment other than surgery /laser; diabetes ; Human Immunodeficiency Virus-positive, immunosuppressed and/or using immunosuppressive therapies; drug abuse.

interventions compared

* Control Placebo nitrite cream and placebo citric acid cream twice daily
* A) 3% sodium nitrite + 4.5% citric acid creams twice daily
* B) 6% sodium nitrite + 9% citric acid creams once daily
* C) 6% sodium nitrite + 9% citric acid creams twice daily

Outcomes

* Primary proportion of patients with complete clearance of target warts Secondary
* Time to clearance
* Wart area
* Wart count
* Patient and investigator assessment of efficacy
* Safety
* Tolerability
* Adherence

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 18 years of age
* 2-50 warts in the anogenital region.
* Female patients of child-bearing potential had to be willing to use a non-barrier method of contraception at entry and for the duration of the study.
* all patients had to be willing to use barrier protection for the duration of the study.
* All patients had to be able to comply with the requirements of the protocol and be likely to return for follow-up visits and had to be contactable for the duration of the study.

Exclusion Criteria:

* Patients with clinically relevant abnormal haematology or biochemistry results (determined from the sample taken at Visit 1).
* Patients who had used an active therapy for anogenital warts within 2 weeks of randomisation to study drug, i.e. Visit 2.
* Patients who had used any local supportive medication, including topical corticosteroids or beta-interferon, within 2 weeks of study entry.
* Patients who had used medication known to adversely affect their haematology profile, including local anaesthetics (benzocaine, lidocaine, etc), nitrofurantoin, sulphonylureas and sulphonamides within 2 weeks of study entry. [Word 'adversely' added by Protocol Amendment 2, 7 May 2002.]
* Patients with abnormal anogenital skin, such as eczema, or skin that had not healed following surgery (cryosurgery, laser ablation or similar).
* Patients who were known to have a concomitant sexually transmitted disease that inhibited accurate assessment of their warts.
* Patients who required treatment other than surgery or laser for internal warts.
* Male patients with intra-urethral warts [deleted by Protocol Amendment 2, 7 May 2002].
* Patients with diabetes (Type I or Type II diabetes).
* Patients who were known to be HIV-positive.
* Patients who were known to be immunosuppressed and/or using immunosuppressive therapies.
* Patients known to abuse alcohol and/or drugs or with a history of chronic alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2001-09; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete clearance of target warts in Intention to treat (ITT) population | 24 weeks
  * Number of and area of target warts (up to 10 selected) at Baseline and Week 1, 2, 4, 6, 8, 10 and 12/withdrawal/early completion and at follow-up (Weeks 4, 8 and 12 after end of treatment)
  * Number of warts at Baseline (Week 0) and of remaining baseline warts at Week 1, 2, 4, 6, 8, 10 and 12/withdrawal/early completion and at Weeks 4, 8 and 12 of follow-up

SECONDARY OUTCOMES:
Total number of warts (baseline and new) at end of treatment | 12 weeks
Patient assessment of efficacy | 12 weeks
  Patient assessment of efficacy (categorised as complete clearance, significant improvement, partial improvement, no change or worsening) at Week 12/withdrawal/early completion
Investigator assessment of efficacy | 12 weeks
  Investigator assessment of efficacy (categorised as complete clearance, significant improvement, partial improvement, no change or worsening) at Week 12/withdrawal/early completion
Patient assessment of tolerability | 12
  Patient assessment of itching, pain and burning (categorised as none, mild, moderate or severe) at treatment site at Screening and Weeks 1, 2, 4, 6, 8, 10 and 12/withdrawal/early completion
Investigator assessment of tolerability | 12 weeks
  Investigator assessment of erythema/eschar and oedema (using modified Draize scales from 0 to 4) at Baseline (Week 0), Weeks 1, 2, 4, 6, 8, 10 and 12/withdrawal/early completion and at follow-up (Weeks 4, 8 and 12 after end of treatment)
Safety of treatment | 12 weeks and followed up
  Adverse events throughout treatment period; unresolved events at end of treatment were followed up Heart rate and blood pressure at each visit during treatment Laboratory tests at Screening and Week 12/withdrawal/early completion Physical examination at Screening and at Week 12/withdrawal/early completion.

OTHER OUTCOMES:
Investigator assessment of staining | 12 weeks
  Investigator assessment of staining (present or absent) at treatment site at Weeks 1, 2, 4, 6, 8, 10 and 12/withdrawal/early completion

CONTACTS AND LOCATIONS:
Overall Officials: Willem I Van der Meijden, Principal Investigator — Erasmus Medical Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ormerod AD, van Voorst Vader PC, Majewski S, Vanscheidt W, Benjamin N, van der Meijden W. Evaluation of the Efficacy, Safety, and Tolerability of 3 Dose Regimens of Topical Sodium Nitrite With Citric Acid in Patients With Anogenital Warts: A Randomized Clinical Trial. JAMA Dermatol. 2015 Aug;151(8):854-61. doi: 10.1001/jamadermatol.2015.0381. PMID 25922903